CLINICAL TRIAL: NCT05901298
Title: Development of 'My Breastfeeding Guide' Mobile Nursing Application and Its Effect on Breastfeeding Process, Self-Efficacy, Infant Nutrition and Attachment
Brief Title: Development of 'My Breastfeeding Guide' Mobile Nursing Application
Acronym: Nursing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Emine Temizkan Sekizler, Lecturer, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SBF-HB-ETS-01
Record Dates: First submitted 2023-05-16; First posted 2023-06-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Self Efficacy; Breast Feeding; Attachment
Keywords: Breastfeeding; Nurse; Mobile application; Self-efficiency
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: The research will be designed in two groups as the mobile nursing practice group (intervention) developed based on Dennis's Breastfeeding Self-Efficacy Theory and Pender's Health Promotion Model and standard care group (control).
Who Masked: Outcomes Assessor
Masking Description: Simple random sample selection will be made using the 'www.randomizer.org' program, and the pregnant women who accepted to participate in the study will be divided into intervention and control groups. To ensure randomization; Age, education level and number of births will be matched. The research will be designed in two groups as the mobile nursing practice group (intervention) and standard care group (control). In the study "The sample size was calculated at the 95% confidence level by using the "G. Power-3.1.9.2" program. As a result of the analysis, with considering the data loss, 10 people will be added to the groups and 44 people will be reached for the intervention group and 44 for the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Application (Experimental): "My Breastfeeding Guide" mobile nursing application, which was developed based on Dennis' Breastfeeding Self-Efficacy Theory and Pender's Health Promotion Model.
  Interventions: Device: My Breastfeeding Guide
- Standart Care (No Intervention): Standard antenatal and postnatal care from health care providers.

INTERVENTIONS:
Device: My Breastfeeding Guide — Development of the content of the mobile nursing application had began with a literature review on breastfeeding, Dennis' Breastfeeding Self-Efficacy Theory and Pender's Health Promotion Model and after content is created. The mobile nursing application can be download via the Google Play Store® and the Apple Store®. The application consist of three parts. In the first part includes mother and baby information which is asked with scales and forms, the second part includes literature knowledge and the third section includes the expert consultation and blog section. Mothers receive notifications consisting of sentences every two days to increase their breastfeeding self-efficacy. The application web page can allow the mothers' information to be kept in the system.
  Arms: Mobile Application

SUMMARY:
The research was planned to develop the "My Breastfeeding Guide" mobile nursing application, which was developed based on Dennis' Breastfeeding Self-Efficacy Theory and Pender's Health Promotion Model, and to determine its effect on the postpartum breastfeeding process, breastfeeding self-efficacy, infant feeding and attachment. The research is in randomized controlled experimental and longitudinal (prospective) design. The research will be carried out with pregnant women who applied to Famagusta State Hospital Obstetrics and Gynecology Polyclinic and a pregnant polyclinic of a private hospital in Famagusta. Pregnant women who applied to Famagusta State Hospital Gynecology and Obstetrics Polyclinic and private hospital's pregnancy polyclinic and met the inclusion criteria of the study will constitute the population of the research. The research will be designed in two groups as the mobile nursing practice group (intervention) and standard care group (control) developed based on Dennis's Breastfeeding Self-Efficacy Theory and Pender's Health Promotion Model. By calculating the sample size in the research, 44 people in the intervention group and 44 people in the control group will reach a total of 88 people. Pregnant Identification Form, Maternal Information Form, Breastfeeding Self-Efficacy Short Form Scale (Postnatal Form), Antenatal Self-Efficacy Short Form Scale, Infant Nutrition Attitude Scale, Breastfeeding Rating Scale, Maternal Attachment Scale and Breastfeeding Self-assessment Form will be used to collect data. Statistical analyzes of the data obtained from the research will be made using the Statistical Package for the Social Science (SPSS) 20.0 package program. While evaluating the research data, frequency, percentage, mean, standard deviation, median, variance analysis from descriptive statistical methods will be used. For homogeneity test between intervention and control groups, the Chi-square test for categorical variables, Mann Whitney test for numerical variables, and sociodemographic variables (age, education status, employment status of himself and his spouse, income level, etc.) and whether the groups are similar in terms of some characteristics. U test will be used. The conformity of the scale scores to the normal distribution will be evaluated with the Shapiro-Wilk test. The results will be evaluated at the 95% confidence level, and the significance at the p<0.05 level.

DETAILED DESCRIPTION:
Aim:

The research was planned to develop the "My Breastfeeding Guide" mobile nursing application, which was developed based on Dennis' Breastfeeding Self-Efficacy Theory and Pender's Health Promotion Model, and to determine its effect on the postpartum breastfeeding process, breastfeeding self-efficacy, infant feeding and attachment.

Hypotheses:

1. H1: Postpartum breastfeeding self-efficacy score averages of the intervention group using the mobile nursing application developed based on the model are higher than the control group.
2. H1: Postpartum infant feeding attitude mean score of the intervention group using the mobile nursing application developed based on the model is higher than the control group.
3. H1: Postpartum breastfeeding mean score of the intervention group using the mobile nursing application developed based on the model is higher than the control group.
4. H1: Postpartum maternal-newborn attachment point averages of the intervention group using the mobile nursing application developed based on the model are higher than the control group.

Type of Research:

It is a randomized controlled experimental and longitudinal (prospective) study.

Place and Time of Research:

The research will be carried out with pregnant women who applied to Famagusta State Hospital Obstetrics and Gynecology Polyclinic and a pregnant polyclinic of a private hospital in Famagusta. The care services of both hospitals are limited to the hospital. Following the approval of the research ethics committee, data collection, data analysis and preparation of the research report are planned as twenty-four months (September 2022-September 2024).

Pilot (preliminary) research:

Pilot (preliminary) research is the preliminary version of the main research and is carried out to determine the feasibility of the main research and the difficulties in conducting the research. Four people will be recruited for each group to represent 10% of the people included in the sample for the pilot (preliminary) study. The purpose of the study was explained to each pregnant woman who was included in the pilot application and their written consent was obtained. The obtained data were analyzed using statistics and it was determined that the research was applicable. Therefore, it was decided to continue the research without making any changes. Mothers in the pilot study were also included in the main study.

Collection of Research Data:

Breastfeeding counseling to be implemented will be carried out in line with the TR Ministry of Health Postpartum Care Management Guide, WHO, UNICEF recommendations for successful breastfeeding, since there is no protocol for prenatal and postnatal care in the TRNC, and the collection of research data starts in the prenatal period and continues in the postpartum period. will continue.

The data will be collected by the researcher from pregnant women who applied to the Famagusta State Hospital Obstetrics and Gynecology Polyclinic and a pregnant outpatient clinic of a private hospital in Famagusta, who met the inclusion criteria and accepted to participate in the study. After the follow-ups in the polyclinic, the pregnant women will be directed to the Breastfeeding Polyclinic where the researcher is located. Pregnant women will be informed about the purpose and process of the research, and pregnant women who volunteered to participate in the research will be evaluated according to the criteria for inclusion in the research. Randomization will be made for those who meet the criteria for inclusion in the study, and after the intervention and control groups are determined, informed consent form and written consent will be obtained. After the implementation of the data collection tools, the intervention and control groups will be trained using the Breastfeeding Education Booklet and a Breastfeeding Education Brochure will be given as a summary of the training. Afterwards, pregnant women in the intervention group will be asked to download and follow the mobile nursing application on their phones throughout the duration of the research.

After the first encounter with the pregnant woman, other data will be collected at 24 for postpartum vaginal deliveries, at 48 hours for cesarean deliveries, at one week, at six weeks, and at six months. At the specified follow-up times, while the intervention group fills in the data collection tools via the mobile nursing application, the mothers in the control group will be contacted via Whatsapp and asked to fill them out via Google Forms®. To avoid data loss, each question will have to be answered and each form will be allowed to be filled once to avoid duplication.

Pregnancy identification form at the first encounter with the pregnant woman, AEÖS to identify mothers with a high risk of stopping breastfeeding prematurely and giving additional food, BBQ to measure breastfeeding attitudes regarding issues such as initiation and maintenance of breastfeeding, approach to formula use, 24 for postpartum vaginal deliveries, cesarean section deliveries In the first 48 hours, the mother's identification form for the mother in the first 48 hours, the EAS to determine how competent the mothers feel about breastfeeding, the IBFAT to evaluate the limitations of breastfeeding in the early postpartum period, and the Breastfeeding Self-Assessment Form for the mother in the intervention group to evaluate her own breastfeeding, the mother at the first week postpartum. Introductory form, EÖÖ, IBFAT and Breastfeeding Self-Assessment Form for the same reasons, mother identification form at the sixth week postpartum, EÖÖ, IBFAT, Breastfeeding Self-Assessment Form for the same reasons, and MDS due to the attachment phase for six to eight weeks after birth. In order to find out whether breastfeeding is continued in the last month, the mother's introduction form, the EÖÖ and the Breastfeeding Self-Assessment Form will be applied for the mother to evaluate her own breastfeeding.

Breastfeeding Education Booklet:

Education with the breastfeeding education booklet will be applied to both the intervention and control groups at the time of the first encounter with the pregnant women, after the application of the data collection tools. The booklet will be developed based on Dennis' Breastfeeding Self-Efficacy Theory and Pender's Health Promotion Model. Since there is no antenatal and postnatal care guide published by the TRNC Ministry of Health, the Turkish Ministry of Health Antenatal Care Management Guide and Postpartum Care Management Guide are eight sub-titles of WHO and UNICEF's ten step recommendations for successful breastfeeding. It has been prepared in line with basic clinical practice recommendations. The recommendations are as follows (WHO, 2018);

1. Pregnant women and their families are informed about the importance and management of breastfeeding.
2. Mothers are provided with skin-to-skin contact with their babies as soon as they are born, and mothers are supported to start breastfeeding as soon as possible and to maintain uninterrupted contact.
3. Support is offered to mothers in initiating and maintaining breastfeeding and managing common difficulties.
4. Unless there is a medical necessity, any food or liquid other than breast milk is not given to the newborn.
5. It is ensured that mothers are kept together with their babies and stay in the same room 24 hours a day.
6. Mothers are supported in recognizing and responding to the signs their babies give when their babies are hungry.
7. Counseling services are provided to mothers on bottle and pacifier use and its risks.
8. Before discharge, parents and their babies are informed about the centers where they will be able to access continuous support and care services for breastfeeding.

In this direction, the aim of the breastfeeding education booklet is to develop and maintain the right breastfeeding behavior in the long term, and therefore to improve breastfeeding rates in the first six months and after, by providing information on the importance and application of breast milk and breastfeeding. After the content of the booklet was created, expert opinion was taken to evaluate it in terms of literacy, intelligibility, relevance and cultural suitability. For this purpose, the content was delivered electronically to 10 faculty members in the field of Women's Health and Diseases Nursing. The final version of the content of the booklet was created in line with the changes suggested for the content in line with the expert opinions.

In order to ensure the content validity of the booklet, the opinion of an expert group consisting of 10 experts in the field was sought. Davis Method was used in the evaluation of expert opinions. According to this method, 1-4 ((1) Unsuitable, (2) Item needs to be corrected appropriately, (3) Applicable but needs minor modification, (4) Very appropriate) were applied for each item. As a result of the opinions obtained, the Content Validity Index of all the titles that make up the booklet was calculated. The criterion value for the Scope Validity Index is accepted as 0.80 and the minimum validity rate for each item should be 0.80. According to the results, the content validity index of all items is 0.80 and above.

Breastfeeding Education Leaflet:

The breastfeeding education brochure will be applied to both the intervention and control groups at the time of first encounter with the pregnant women, after the application of the data collection tools and the breastfeeding education booklet. The brochure will be developed based on Dennis' Breastfeeding Self-Efficacy Theory and Pender's Health Promotion Model. Since there is no antenatal and postnatal care guide published by the TRNC Ministry of Health, the TR Ministry of Health Antenatal Care Management Guide and Postpartum Care Management Guide, WHO and UNICEF's ten step recommendations for successful breastfeeding are eight basic clinical practices. will be prepared in accordance with the recommendations. After the content of the brochure was created, expert opinion was taken to evaluate it in terms of literacy, intelligibility, relevance and cultural suitability. For this purpose, the content was delivered electronically to 10 faculty members in the field of Women's Health and Diseases Nursing. In line with the expert opinions, the final version of the brochure content was created in line with the changes suggested for the content.

In order to ensure the content validity of the brochure, the opinion of an expert group consisting of 10 experts in the field was sought. Davis Method was used in the evaluation of expert opinions. According to this method, 1-4 ((1) Unsuitable, (2) Item needs to be corrected appropriately, (3) Applicable but needs minor modification, (4) Very appropriate) were applied for each item. As a result of the opinions obtained, the Scope Validity Index was calculated for all the items that make up the brochure section content. The criterion value for the Scope Validity Index is accepted as 0.80 and the minimum validity rate for each item should be 0.80. According to the results, the content validity index of all items is 0.80 and above.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 and over,
* Women who are in the last trimester of pregnancy (32nd gestational week and above),
* Women with singleton pregnancy,
* Women who do not have any health problems that may prevent breastfeeding,
* Women with smartphones with Android and iOS operating systems,
* Women who can access the Internet,
* There will be women who do not have literacy problems, mental disabilities and communication problems.

Exclusion Criteria:

* Women under 18 years of age,
* Women who are under the last trimester of pregnancy (32nd week of pregnancy),
* Women who do not speak Turkish,
* Women who own a smartphone with an operating system other than Android and iOS.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Pregnant Introduction Form | Between 32nd - 42nd gestational week
  The Pregnant Introductory Form was created by the researcher using the literature. The form contains personal information and pregnancy information.
Mother Introductory Form | Postpartum first 24-48 hours,1st-6th week, 6th month
  The Mother Identification Form was created by the researcher using the literature. Form consists of a total of 15 questions, such as including information such as feeding the baby, giving a pacifier to the baby, giving a bottle to the baby, breastfeeding frequency in the first 24 hours.
Breastfeeding Self-Efficacy Short Form Scale (Postnatal Form) | Postpartum first 24-48 hours,1st-6th week, 6th month
  The Breastfeeding Self-Efficacy Scale was developed to evaluate the breastfeeding self-efficacy levels of mothers. The lowest score that can be obtained from the scale is 14, and the highest score is 70. A high score indicates that breastfeeding self-efficacy is high.
Antenatal Self-Efficacy Short Form Scale | Between 32nd - 42nd gestational week
  Antenatal Self-Efficacy Short Form Scale was developed to evaluate the breastfeeding self-efficacy levels of mothers in antenatal period. The lowest score that can be obtained from the scale is 14, and the highest score is 70. A high score indicates that breastfeeding self-efficacy is high.
Infant Nutrition Attitude Scale (BBTS) | Between 32nd - 42nd gestational week
  The Iowa Infant Feeding Attitude Scale (Iowa Infant Feeding Attitude Scale) evaluates women's attitudes towards breastfeeding and to predict breastfeeding duration as well as the choice of infant feeding method. The total attitude score ranges from 17 (reflecting a positive attitude in bottle feeding) to 85 points (reflecting a positive attitude in breastfeeding).
Breastfeeding Rating Scale (IBFAT) | Postpartum first 24-48 hours,1st-6th week
  The Infant Breastfeeding Assesment Tool (IBFAT) evaluates the limitations of breastfeeding adequacy at each feeding, and the Turkish validity and reliability of the scale was performed by Çelik and Demirci in 2017. The scale consists of six questions and scores are made based on the answers of the mothers to the questions. Each question is evaluated between 0-3 points and the highest score is 12. The score range for effectively fed infants is 10-12 points.
Maternal Attachment Scale | Postpartum 6th week
  The Maternal Attachment Scale (MBI) is a 26-item, four-point Likert-type scale developed by Mary E. Muller in 1994 to measure attachment with maternal love. Turkish validity and reliability of the scale was done by Kavlak and Şirin in 2009. The lowest score that can be obtained from the scale is 26, and the highest score is 104. A high score indicates high maternal attachment. It is recommended to apply the scale to mothers who have babies between one and four months postpartum.
Breastfeeding Self-Assessment Form | Postpartum first 24-48 hours,1st-6th week, 6th month
  The Breastfeeding Self-Assessment Form was created by the researchers on the basis of the Turkish Ministry of Health Breastfeeding Observation Form, in order for the mothers in the intervention group to evaluate their breastfeeding through the 'My Breastfeeding Guide' mobile nursing application. The form includes body position, baby's behavior, time spent sucking and sucking. This form does not have a scoring system. The purpose of using the form is for mothers to evaluate their own breastfeeding while using the mobile application.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Doan TTD, Tran TC, Pham NM, Zhao Y, Dinh TPH, Hoai NX, Lee A, Binns C, Bui TTH. Designing and developing a mobile app (BeBo) in a randomized controlled trial study to promote breastfeeding among Vietnamese mothers. Int Breastfeed J. 2023 Jan 19;18(1):7. doi: 10.1186/s13006-023-00543-7. PMID 36658643
- [Result] Lewkowitz AK, Lopez JD, Carter EB, Duckham H, Strickland T, Macones GA, Cahill AG. Impact of a novel smartphone application on low-income, first-time mothers' breastfeeding rates: a randomized controlled trial. Am J Obstet Gynecol MFM. 2020 Aug;2(3):100143. doi: 10.1016/j.ajogmf.2020.100143. Epub 2020 May 17. PMID 33345878
- [Result] Meedya S, Win K, Yeatman H, Fahy K, Walton K, Burgess L, McGregor D, Shojaei P, Wheatley E, Halcomb E. Developing and testing a mobile application for breastfeeding support: The Milky Way application. Women Birth. 2021 Mar;34(2):e196-e203. doi: 10.1016/j.wombi.2020.02.006. Epub 2020 Feb 17. PMID 32081557